CLINICAL TRIAL: NCT04773119
Title: AF Burden and Echo-guided Persistent AF Ablation Strategy Using Either PV Isolation Alone (CLOSE Protocol) or Optimized Compartmentalization of the Left Atrium (Pseudo-maze Technique): the CLOSEMAZE Study
Brief Title: AF Burden and Echo-guided Persistent AF Ablation Strategy Using Either PV Isolation Alone (CLOSE Protocol) or Optimized Compartmentalization of the Left Atrium (Pseudo-maze Technique)
Acronym: CLOSEMAZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Sebastien Knecht, Principal Investigator, AZ Sint-Jan AV
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2312
Record Dates: First submitted 2021-02-10; First posted 2021-02-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulmonary vein isolation (PVI) only (Active Comparator)
  Interventions: Procedure: PVI only
- PVI with substrate (Active Comparator)
  Interventions: Procedure: PVI with substrate ablation

INTERVENTIONS:
Procedure: PVI only — Patients in this group receive PVI only
  Arms: Pulmonary vein isolation (PVI) only
Procedure: PVI with substrate ablation — Patients in this group receive PVI as well as substrate ablation
  Arms: PVI with substrate

SUMMARY:
Recent publications suggest that neither empirical nor individualized substrate modification strategies could improve single-procedure efficacy beyond pulmonary vein (PV) isolation for persistent atrial fibrillation (AF). However, persistent AF represent a broad spectrum of the same disease and if PV isolation may be sufficient for some patient with self-terminated AF or with a small left atrium, a more extended substrate ablation may be required for other patients, for which a second procedure for atrial tachycardia (AT) recurrence is then frequently needed. In addition, a lot of progress has recently been made in the field of ablation techniques using contiguous and optimized ablation radiofrequency (RF) lesions and also for AT mapping with promising results using repetitive but discontinuous Holter monitoring.

This trial aims at

1. To objectively compare atrial tachyarrhythmia (ATA) burden > 2 months before ablation and after one or two 'CLOSEMAZE'-guided ablation(s) using continuous monitoring and echo data as a guide for the ablation strategy during the first ablation.
2. To assess ATA burden using continuous monitoring up to 3 years after ablation.
3. To identify baseline structural and electrical properties of the atria or procedural characteristics that predict 1-year and 3-year outcome.

ELIGIBILITY:
Inclusion Criteria

1. Patients with symptomatic persistent AF (history of continuous AF > 7 days), meeting following criteria at the out-patient clinic:

   * patient has AF at the time of the visit
   * AF episodes are symptomatic, and patient is drug-resistant (at least one class Ic or III), or drug-intolerant (palpitations, fatigue, dyspnea, cardiomyopathy,…)
   * If the patient has heart failure (LVEF<50%), first line AF ablation (instead of amiodarone) is indicated
2. Signed Patient Informed Consent Form.
3. Age 18 years or older.
4. Able and willing to comply with all follow-up testing and requirements.

Exclusion Criteria

1. Longstanding persistent atrial fibrillation (Suspected continuous AF>1 year)
2. Previous ablation for AF
3. left atrial antero-posterior diameter > 55 mm (parasternal long axis view (PLAX))
4. LVEF < 30% (ejection fraction)
5. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
6. Coronary artery bypass graft within the last three months
7. Awaiting cardiac transplantation or other cardiac surgery
8. Documented left atrial thrombus on imaging
9. Diagnosed atrial myxoma
10. Women who are pregnant or breastfeeding
11. Acute illness or active systemic infection or sepsis
12. Unstable angina
13. Uncontrolled heart failure
14. Myocardial infarction within the previous two months
15. History of blood clotting or bleeding abnormalities
16. Contraindication to anticoagulation therapy (ie, heparin or warfarin)
17. Life expectancy less than 12 months
18. Enrollment in any other study evaluating another device or drug
19. Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Atrial tachyarrhythmia (ATA) burden before and after 'CLOSEMAZE'-guided based ablation and off anti-arrhythmic drug (AAD) therapy | CLR implant to 3 year post ablation
  ATA burden (= time that a subject experiences AF) will be monitored with continuous loop recording (CLR) from time of CLR implant until 3 years after ablation

SECONDARY OUTCOMES:
Atrial tachyarrhythmia burden after one CLOSEMAZE guided ablation | 3 years after ablation
  ATA burden after first ablation documented through continuous loop recordings
Atrial tachyarrhythmia burden after two CLOSEMAZE guided ablation | 3 years after ablation
  ATA burden after two ablations documented through continuous loop recordings

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Knecht, MD, PhD, Principal Investigator — AZ Sint-Jan AV
Locations (1):
- AZ Sint-Jan Brugge-Oostende AV, Bruges, West-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No